CLINICAL TRIAL: NCT05046015
Title: Comparing Dry to Very Dry and Cracked Foot Skin Between Diabetic and Non-diabetic Subjects and the Effects of Two Cosmetic leave-on Foot Products: an Exploratory Study
Brief Title: Comparison Dry Foot Skin Between Diabetic and Non-diabetic Subjects and the Effects of Two Cosmetic Foot Care Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.109799
Record Dates: First submitted 2020-07-29; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2017-02

CONDITIONS: Xerosis Cutis
Keywords: Diabetes type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Single Blind (Investigator) Non-Randomized 60 [Anticipated]
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non diabetic (No Intervention): Control Group of 20 non-diabetics. Skin measurements, evaluation of skin dryness and sampling of skin particles will be performed
- moderate dryness-diabetic (Experimental): Experimental: Diabetics with moderate dryness. Intervention Group of 20 diabetics with moderate dryness
  10% Urea foot lotion During the course of the study participants cleanse one foot (previously randomized) once daily using the mild cleanser "Cetaphil® Restoraderm Body Wash" and apply the product "Excipial® U10 Lipolotion 10% Urea" once daily in the evening by themselves.
  Interventions: Other: 10% Urea foot lotion
- severe dryness- diabetic (Experimental): Intervention Group of 20 diabetics with severe dryness 10% Urea foot ointment During the course of the study participants cleanse their feet once daily using the mild cleanser "Cetaphil® Restoraderm Body Wash" and apply the product "Excipial® Fuss Salbe 10% Urea" on both feet once daily in the evening by themselves.
  Interventions: Other: 10% Urea foot ointment

INTERVENTIONS:
Other: 10% Urea foot lotion — During the course of the study participants cleanse one foot (previously randomized) once daily using the mild cleanser "Cetaphil® Restoraderm Body Wash" and apply the product "Excipial® U10 Lipolotion 10% Urea" once daily in the evening by themselves.
  Arms: moderate dryness-diabetic
Other: 10% Urea foot ointment — During the course of the study participants cleanse one foot (previously randomized) once daily using the mild cleanser "Cetaphil® Restoraderm Body Wash" and apply the product "Excipial® U10 ointment10% Urea" once daily in the evening by themselves.
  Arms: severe dryness- diabetic

SUMMARY:
The overall aims of this study are to compare the structure and function of dry to very dry and cracked foot skin between diabetic and nondiabetic subjects and to evaluate the effects of two cosmetic leave-on products on dry and fissured diabetic foot skin.

Specific issues are:

Are there any differences between the morphological and functional characteristics of dry to very dry and cracked skin foot between diabetic and nondiabetic subjects? What are the effects of a 4-week once daily application of an intensive care foot ointment (urea 10% foot ointment) or foot lotion (10% Urea foot lotion) on the skin barrier and on clinical signs of dryness and fissures?

DETAILED DESCRIPTION:
A long existing diabetes mellitus type II is often associated with a number of skin changes. Xerosis Cutis is the most common skin alteration. The risk of diabetics of developing a foot ulcer is estimated to be 15%. Very dry and cracked skin represents an additional risk factor, so that adequate skin care is a widely recommended intervention in diabetic patients. But there are only few studies investigating the skin barrier structure and function in diabetic patients. Available study results seem to suggest, that for instance sebum content, stratum corneum hydration, and pH are associated with Diabetes mellitus.

The overall aims of this study are to compare the structure and function of dry to very dry and cracked foot skin between diabetic and nondiabetic subjects and to evaluate the effects of two cosmetic leave-on products on dry and fissured diabetic foot skin.

Specific issues are:

Are there any differences between the morphological and functional characteristics of dry to very dry and cracked skin foot between diabetic and nondiabetic subjects? What are the effects of a 4-week once daily application of an intensive care foot ointment (urea 10% foot ointment) or foot lotion (10% Urea foot lotion) on the skin barrier and on clinical signs of dryness and fissures?

ELIGIBILITY:
diabetics and non-diabetics

* Age 40 to 75 years
* Moderate (categories 3 and 4), severe (category 5) dry skin according to the classification of Rogers et al. 1989
* Degree of dryness comparable on both feet (maximum 1 category difference)
* BMI between 18.5 and 34.9 kg/m2 (normal weight to class I obesity)
* Able to understand and comply with the study requirements
* additionally only for diabetics: Diabetes mellitus type 2 for at least 3 years according to Patient

Exclusion Criteria:

* diabetics and non-diabetics
* Any kind of adverse foot condition except xerosis like nail injury, ulceration, (suspected) infection including fungal infection
* History of adverse foot condition except xerosis and tinea pedis, like nail injury, ulceration, pain
* Mild xerosis cutis of feet (categories 1 and 2 according to Rogers et al. 1989)
* Severe xerosis cutis of feet (category 6 according to Rogers et al. 1989)
* Gait problems
* Other non-controlled chronic and/or acute skin disease except xerosis (e.g. atopic dermatitis, psoriasis, tinea pedis)
* Unstable chronic systemic disease (e.g. hypertension, renal insufficiency)
* Acute systemic disease (e.g. infection)
* Body temperature > 38°C
* Pain anywhere
* Wear of compression stockings at any time
* Use of topical steroids
* Use of skin care leave-on products on the feet in the previous 2 weeks
* Known hypersensitivity or allergy to product ingredients
* Drugs that might affect sweating (oral corticosteroids, psychoactive drugs)
* Topical treatments other than the study products on the test areas within14 days prior Day 0 and during the course of the study
* Pedicure/ medical foot care 14 days prior D 0 and during the course of the study
* Any condition/ circumstance (e.g. cognitive impairment, visual impairment) that might interfere with study compliance in the opinion of the investigator
* Current participation in another clinical study
* Subject is institutionalized because of legal or regulatory order
* additionally only for non-diabetics: Diabetes mellitus type 2 according to Patient
* additionally only for diabetics:
* Charcot osteoarthropathy
* Neuropathy tested with a Semmes-Weinstein monofilament (according to Bakker et al. 2012)
* Absence of pedal pulses (1) Posterior tibial artery (2) Dorsalis pedis artery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Overall Dry Skin Score | Baseline; Day 28±2
  Clinical assessment of the presence or severity of skin dryness using a 7 point scale at the sole of the foot (randomized). A score of '0' indicated normal skin/no sign of dryness, whereas a score of '6' indicates large-scale plates, deep erythematous fissures and cracks

SECONDARY OUTCOMES:
Skin barrier | Day 0, Day 14±1,Day 28±2
  Transepidermal water loss: Measurement using the Tewameter®
  Three replicate measurements; according to the Technical Procedures G01_A1_V01 g/m2/h

OTHER OUTCOMES:
Stratum corneum hydration | Day 28
  Stratum corneum hydration - Measurement using the Corneometer at Day 28
Skin surface pH | Day 0 , Day 14, Day 28
  Skin surface pH
  Measurement using the pH-Meter® Three replicate measurements; according to the Technical Procedures G01_A4_V01
Epidermal thickness | D28
  Epidermal thickness
  Measurement using OCT taking one image/ visit/ test area Mean of three epidermal thickness measurements; according to the Technical Procedures G04_A1_V01 μm
Skin surface topography | Day 0, Day 28±2
  Skin surface topography - Measurement using Visioscan®
Elasticity/Stiffness | Day 28
  Elasticity/Stiffness Measurement using Cutometer® at day 28
lipids | Day 0, Day 28
  Oxidative stress on lipids Measurement according to sampling method of Synelvia (Version 2)
Callus | Day 0, Day 28
  Callus
  * Clinical evaluation by study investigator
  * Classification of Callus severity according to Hashmi et al. 2015
Cracks/ Fissures | Day 0, Day 28
  Cracks/ Fissures
  * Clinical evaluation by study investigator
  * Classification according to Oe et al. 2012

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Blume -Peytavi, Prof Dr.med, Principal Investigator — Charité Universitatsmedizin Berlin; Ulrike Blume-Peytavi, Prof Dr.med, Principal Investigator — Charité Universitatsmedizin Berlin
Locations (1):
- Charité Universitatsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No